CLINICAL TRIAL: NCT06310824
Title: A Randomized, Double-blind, Controlled, Parallel-group, Single Dose, Three-arm Study to Compare the Pharmacokinetic Similarity of MAB-22 Versus Prolia® Sourced From the European Union and United States in Healthy Male Participants
Brief Title: Single Dose, Three-arm Study to Compare the Pharmacokinetic Similarity of MAB-22 Versus Prolia®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xentria, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MAB-22-101
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MAB-22 (Experimental): Single subcutaneous injection on Day 1
  Interventions: Drug: MAB-22
- EU-Prolia® (Active Comparator): Single subcutaneous injection on Day 1
  Interventions: Drug: EU-Prolia®
- US-Prolia® (Active Comparator): Single subcutaneous injection on Day 1
  Interventions: Drug: US-Prolia®

INTERVENTIONS:
Drug: MAB-22 — 60mg dose of a single subcutaneous injection
  Arms: MAB-22
Drug: EU-Prolia® — 60mg dose of a single subcutaneous injection
  Arms: EU-Prolia®
Drug: US-Prolia® — 60mg dose of a single subcutaneous injection
  Arms: US-Prolia®

SUMMARY:
A Randomized, Double-blind, Controlled, Parallel-group, Single Dose, Three-arm Study to Compare the Pharmacokinetic Similarity of MAB-22 Versus Prolia®

DETAILED DESCRIPTION:
This study is a Phase 1, double-blind, randomized, single dose, parallel-group, 3-arm, Pharmacokinetic (PK) study designed to assess the biosimilarity, including the PK, Pharmacodynamics (PD), safety, tolerability, and immunogenicity of MAB-22 compared with reference Prolia® sourced from the European Union (EU) and United States (US) after single subcutaneous (SC) injection in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male participants between 25 and 55 years of age (inclusive) on the day of signing the informed consent.
2. Have a body weight between 50.0 and 110.0 kg (inclusive) and a body mass index (BMI) between 18.0 and 32.9 kg/m2 (inclusive).
3. Have 12-lead electrocardiogram (ECG) results without clinically significant abnormal findings confirmed by the investigator.
4. Have vital sign results without clinically significant abnormal findings confirmed by the investigator, including but not limited to:

   1. Resting supine systolic blood pressure <145 mmHg and diastolic blood pressure of <90 mmHg.
   2. Heart rate 40 to 100 beats per minute (bpm).
   3. Respiration rate 8 to 20 resp/min.
   4. Temporal or ear temperature 35.5 to 37.6°C.
   5. Oxygen saturation 95 to 100%.
5. Have physical examination results without clinically significant abnormal findings confirmed by the investigator.

Exclusion Criteria:

1. Prior diagnosis of bone disease, or any condition that will affect bone metabolism such as, but not limited to: osteoporosis, osteogenesis imperfecta, hyperparathyroidism, hyperthyroidism, hypothyroidism, osteomalacia, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, current flare-up of osteoarthritis and/or gout, active malignancy, moderate to severe renal disease (defined as glomerular filtration rate <60 mL/min), Paget's disease of the bone, recent bone fracture (within 6 months), or malabsorption syndrome.
2. Osteonecrosis of the jaw (ONJ) or risk factors for ONJ, such as invasive dental procedures (e.g., tooth extraction, dental implants, oral surgery in the past 6 months), poor oral hygiene, periodontal, and/or preexisting dental disease at the determination of the investigator.
3. Recent tooth extraction (within 6 months of the screening visit). Edentulous participants are permitted to enroll in the study, as long as the most recent tooth extraction occurred >6 months prior to the screening visit.
4. Evidence of hypocalcemia (total calcium below the normal range [8.5 to 10.5 mg/dL or 2.21 to 2.65 mmol/L]) at screening.
5. Known vitamin D deficiency (defined as vitamin D <12 ng/mL or <30.0 nmol/L); or known intolerance to calcium or vitamin D supplements. Retest of vitamin D is allowed once. Vitamin D repletion is permitted (e.g., vitamin D supplements) with a tolerable upper intake level of 100 mcg (4000 IU) daily, at the discretion of the investigator.

Ages: 25 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 225 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-07-22 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 extrapolated to infinity (AUC0-∞) | Day 1 to Week 37
  Primary endpoints are to compare Pharmacokinetics (PK) similarity in healthy male participants assessments collected during predose and postdose (Day 1) at 4 and 24 hours, and at Days 3, 7, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253. PK and Pharmacodynamic (PD)
Maximum observed serum concentration (Cmax) | Day 1 to Week 37
  Primary endpoints are to compare Pharmacokinetics (PK) similarity in healthy male participants assessments collected during predose and postdose (Day 1) at 4 and 24 hours, and at Days 3, 7, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253. PK and Pharmacodynamic (PD)

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to the last quantifiable concentration (AUC0-last) | Day 1 to Week 37
  Secondary endpoints are to assess the safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamic (PD), and immunogenicity of MAB-22 versus Prolia® (US-licensed) and Prolia® (EU-approved) in healthy participants assessments collected during predose and postdose (Day 1) at 4 and 24 hours, and at Days 3, 7, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253.
Area under the concentration-time curve | 0 to Week 21
  Secondary endpoints are to assess the safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamic (PD), and immunogenicity of MAB-22 versus Prolia® (US-licensed) and Prolia® (EU-approved) in healthy participants assessments collected during predose and postdose (Day 1) at 4 and 24 hours, and at Days 3, 7, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253.
Area under the concentration-time curve | Week 21 to Week 37
  Secondary endpoints are to assess the safety, tolerability, Pharmacokinetics (PK) and Pharmacodynamic (PD), and immunogenicity of MAB-22 versus Prolia® (US-licensed) and Prolia® (EU-approved) in healthy participants assessments collected during predose and postdose (Day 1) at 4 and 24 hours, and at Days 3, 7, 11, 15, 22, 29, 43, 57, 71, 85, 113, 141, 169, 197, 225, and 253.

CONTACTS AND LOCATIONS:
Locations (2):
- Xentria Investigative Site, Budapest, Hungary
- Xentria Investigative Site, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No